CLINICAL TRIAL: NCT05199038
Title: Comparison of 2 Days Versus 5 Days of Octreotide After Endoscopic Therapy in Preventing Early Esophageal Varices Rebleed: A Randomized Controlled Study
Brief Title: Comparison of 2 Days Versus 5 Days of Octreotide After Endoscopic Therapy in Preventing Early Esophageal Varices Rebleed : A Randomized Controlled Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mennat-Allah Mohammed El Sawaf, melsawaf, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Esophageal Varices Rebleeding
Record Dates: First submitted 2021-12-22; First posted 2022-01-20 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Esophageal Varices
MeSH Terms: conditions — Esophageal and Gastric Varices | interventions — Octreotide

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2 Days of octreotide infusion (Experimental)
  Interventions: Drug: Octreotide
- 5 Days of octreotide infusion (Active Comparator)
  Interventions: Drug: Octreotide

INTERVENTIONS:
Drug: Octreotide — Octreotide infusion for 2 days in patients with bleeding esophageal varices.

SUMMARY:
The aim of this study is to compare the efficacy of 2-days versus 5-days octreotide infusion after endoscopic therapy in preventing early esophageal varices rebleed in patients with cirrhosis.

DETAILED DESCRIPTION:
Variceal hemorrhage, causative of 70% of all upper gastrointestinal (GIT) bleeding events in patients with portal hypertension, remains one of the most severe and immediate life-threatening complications in patients with cirrhosis and constitutes the second most frequent decompensating event after ascites .

Gastro-esophageal varices are identified in about 30% of patients with compensated cirrhosis and 60% of patients with de-compensated cirrhosis . Esophageal variceal bleeding (EVB) occurs in 10-20% of cirrhotic patients per year and each bleeding episode can be associated with in-hospital mortality .

Mortality during the first episode is estimated to 15-20% but is higher in severe patients (Child Pugh C), at around 30%, whereas it is very low in patients with compensated cirrhosis (Child Pugh A) .The main predictors of bleeding in clinical practice are: large versus small varices, red wale marks, Child Pugh C versus Child Pugh A-B .

Treatment of variceal bleeding should be started as soon as bleeding is clinically confirmed, regardless the lack of confirmation by upper endoscopy . Initial therapy should be directed at restoring blood volume. Vasoactive drug therapy and antibiotic prophylaxis should be initiated as soon as AVB is suspected. Goals of therapy in AVB include the control of bleeding, as well as the prevention of early recurrence and the prevention of six-week mortality .

Starting vasoactive drugs before endoscopy decreases the incidence of active bleeding during endoscopy and facilitates endoscopic therapy, improving the control of bleeding, and potentially survival. Terlipressin, somatostatin or octreotide are accepted drugs with proven efficacy .

Once AVB is confirmed, vasoactive drug therapy should be administered for five days to avoid early rebleeding. Shorter administration of vasoactive drugs (48-72 h) can be considered in less severe episodes although more data are required .The optimal duration of pharmacological therapy has not been well established. In randomized-controlled trials, the duration of vasoactive drugs has varied between 8 h and 6 days .

There was a major agreement that an appropriate length of therapy would be anywhere between 2 and 5 days depending on control of hemorrhage and the presence or absence of predictors of rebleeding .

The combination of endoscopic therapy and vasoactive drugs is more effective than the isolated use of either of these options alone, because it combines the local haemostatic effect on the varices induced by endoscopic treatment and the portal hypotensive effect achieved with drugs. This combination is currently considered the standard of care in AVB .

ELIGIBILITY:
Inclusion Criteria:

1. Acute esophageal varices bleeding
2. Liver cirrhosis

Exclusion Criteria:

1. Initial failure to control variceal bleed on endoscopy
2. Other causes of GIT bleeding
3. Hepatocellular carcinoma
4. Portal vein thrombosis
5. Renal dialysis and hepatorenal syndrome
6. History of myocardial infarction
7. Pregnancy or lactation
8. Allergy to octreotide

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Esophageal varices rebleed within 5days after control of initial bleed | with in 5 days after controlof initial bleeding
  5 days Rebleeding means
  1. Recurrence of hematemesis or melena after bleeding control
  2. Sustained tachycardia more than 100 beat/ min and sudden drop of systolic blood pressure less than 100
  3. A drop in hemoglobin by more than 20 percentage points from baseline
  4. Transfusion of >2 unites packed red blood cells after endoscopic intervention of variceal bleeding

SECONDARY OUTCOMES:
Esophageal varices rebleed at 5 days and 6 weeks after control of initial bleed | 5 days - 6 weeks after control of initial bleeding
  5days-6weeks rebleed means
  1. Any new episode of hematemesis, melena, or hematochezia (with sustained tachycardia more than 100 beat/min and drop of systolic blood pressure less than 100)
  2. Drop in hemoglobin by more than 20 percentage points OR the need for >2 units packed red blood cells

REFERENCES:
- [Background] European Association for the Study of the Liver. EASL Clinical Practice Guidelines for the management of patients with decompensated cirrhosis. J Hepatol. 2018 Aug;69(2):406-460. doi: 10.1016/j.jhep.2018.03.024. Epub 2018 Apr 10. No abstract available. PMID 29653741
- [Background] Mallet M, Rudler M, Thabut D. Variceal bleeding in cirrhotic patients. Gastroenterol Rep (Oxf). 2017 Aug;5(3):185-192. doi: 10.1093/gastro/gox024. Epub 2017 Jul 21. PMID 28852523
- [Background] Haq I, Tripathi D. Recent advances in the management of variceal bleeding. Gastroenterol Rep (Oxf). 2017 May;5(2):113-126. doi: 10.1093/gastro/gox007. Epub 2017 Apr 7. PMID 28533909
- [Background] Garcia-Tsao G, Bosch J. Management of varices and variceal hemorrhage in cirrhosis. N Engl J Med. 2010 Mar 4;362(9):823-32. doi: 10.1056/NEJMra0901512. No abstract available. PMID 20200386
- [Background] Seo YS, Park SY, Kim MY, Kim JH, Park JY, Yim HJ, Jang BK, Kim HS, Hahn T, Kim BI, Heo J, An H, Tak WY, Baik SK, Han KH, Hwang JS, Park SH, Cho M, Um SH. Lack of difference among terlipressin, somatostatin, and octreotide in the control of acute gastroesophageal variceal hemorrhage. Hepatology. 2014 Sep;60(3):954-63. doi: 10.1002/hep.27006. Epub 2014 Jul 25. PMID 24415445
- [Background] Azam Z, Hamid S, Jafri W, Salih M, Abbas Z, Abid S, Shah H. Short course adjuvant terlipressin in acute variceal bleeding: a randomized double blind dummy controlled trial. J Hepatol. 2012 Apr;56(4):819-24. doi: 10.1016/j.jhep.2011.11.019. Epub 2011 Dec 16. PMID 22178268
- [Background] Sarin SK, Kumar A, Angus PW, Baijal SS, Baik SK, Bayraktar Y, Chawla YK, Choudhuri G, Chung JW, de Franchis R, de Silva HJ, Garg H, Garg PK, Helmy A, Hou MC, Jafri W, Jia JD, Lau GK, Li CZ, Lui HF, Maruyama H, Pandey CM, Puri AS, Rerknimitr R, Sahni P, Saraya A, Sharma BC, Sharma P, Shiha G, Sollano JD, Wu J, Xu RY, Yachha SK, Zhang C; Asian Pacific Association for the Study of the Liver (APASL) Working Party on Portal Hypertension. Diagnosis and management of acute variceal bleeding: Asian Pacific Association for Study of the Liver recommendations. Hepatol Int. 2011 Jun;5(2):607-24. doi: 10.1007/s12072-010-9236-9. Epub 2011 Feb 19. PMID 21484145
- [Background] Garcia-Tsao G, Sanyal AJ, Grace ND, Carey W; Practice Guidelines Committee of the American Association for the Study of Liver Diseases; Practice Parameters Committee of the American College of Gastroenterology. Prevention and management of gastroesophageal varices and variceal hemorrhage in cirrhosis. Hepatology. 2007 Sep;46(3):922-38. doi: 10.1002/hep.21907. No abstract available. PMID 17879356
- [Background] Villanueva C, Piqueras M, Aracil C, Gomez C, Lopez-Balaguer JM, Gonzalez B, Gallego A, Torras X, Soriano G, Sainz S, Benito S, Balanzo J. A randomized controlled trial comparing ligation and sclerotherapy as emergency endoscopic treatment added to somatostatin in acute variceal bleeding. J Hepatol. 2006 Oct;45(4):560-7. doi: 10.1016/j.jhep.2006.05.016. Epub 2006 Jun 28. PMID 16904224